CLINICAL TRIAL: NCT02502747
Title: RIGENERA 2.0 (Recupero Dall'Infarto Miocardico Con G-CSF E Nuovi Esempi di Rigenerazione Avanzata) Project: "The Combined Effect of Subcutaneous Granulocyte - Colony Stimulating Factor and Myocardial Contrast Echocardiography With Intravenous Infusion of Sulphur Hexafluoride on Post-infarction Left Ventricular Function"
Brief Title: RIGENERA 2.0 Trial
Acronym: RIGENERA
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: slow enrolment
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Principal Investigator, Antonio Maria Leone, MD, MD, PhD, Catholic University of the Sacred Heart
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RIGENERA 2.0
Record Dates: First submitted 2015-06-29; First posted 2015-07-20 (Estimated); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Anterior Myocardial Infarction; Heart Failure
MeSH Terms: conditions — Anterior Wall Myocardial Infarction; Heart Failure

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- G-CSF and Myocardial Contrast Echocardiography (MCE) (Experimental): subcutaneous Granulocyte - Colony Stimulating Factor ( on top of optimal standard of care) and Myocardial Contrast Echocardiography with intravenous infusion of sulphur hexafluoride.
  Interventions: Drug: rhu G-CSF; Procedure: Myocardial Contrast Echocardiography
- Placebo and Myocardial Contrast Echocardiography (MCE) (Active Comparator): Patients will be receive optimal standard of care and Myocardial Contrast Echocardiography with intravenous infusion of sulphur hexafluoride.
  Interventions: Drug: optimal standard of care; Procedure: Myocardial Contrast Echocardiography

INTERVENTIONS:
Drug: rhu G-CSF — rhu G-CSF will be administered 5 µg/kg twice daily for 5 days, subcutaneously
  Other Names: recombinant human Granulocyte - Colony Stimulating Factor
  Arms: G-CSF and Myocardial Contrast Echocardiography (MCE)
Drug: optimal standard of care — Optimal standard of care
  Arms: Placebo and Myocardial Contrast Echocardiography (MCE)
Procedure: Myocardial Contrast Echocardiography — Myocardial Contrast Echocardiography with sulphur hexafluoride.

SUMMARY:
Study Objectives: To determine whether, in patients with large acute myocardial infarction undergoing primary or rescue angioplasty, the administration of subcutaneous Lenograstim [recombinant human Granulocyte-Colony Stimulating Factor (rhu G-CSF), Myelostim 34, Italfarmaco] associated with Myocardial Contrast Echocardiography and the intravenous infusion of sulphur hexafluoride (Sonovue, Bracco) determines an improvement:

* in regional and global contractile function, myocardial perfusion and infarct size assessed by cardiovascular magnetic resonance.
* Echocardiographic parameters of LV function
* in the serum profile of inflammatory and mobilizing cytokines and of biomarkers of myocardial damage and wall stress

DETAILED DESCRIPTION:
1. INTRODUCTION 1.1. BACKGROUND AND RATIONALE OF THE STUDY The long term prognosis of patients suffering from acute myocardial infarction (AMI) has progressively improved since the introduction of reperfusion therapies and in particular primary angioplasty [1]. In the setting of ST-elevation myocardial infarction (STEMI), the immediate reopening of acutely occluded coronary arteries via primary angioplasty is the treatment of choice to salvage ischemic myocardium. However, the sudden re-initiation of blood flow can lead to a local acute inflammatory response with further endothelial and myocardial damage. This phenomenon, described as 'reperfusion injury', may explain why, despite optimum myocardial reperfusion, the short-term mortality after AMI approaches 7% [1] and the incidence of heart failure approaches 15-20% [2][3]. Despite the use of full conventional treatment, including ACE inhibitors, beta-blockers, aldosterone inhibitors and diuretics, in the context of randomised controlled trials yearly mortality rates of patients with post-infarction heart failure are still in the range of 10-13% and rehospitalisation for worsening of heart failure occurs at a yearly rate of 6-8 % [4]. Registry data indicate a more dismal outcome in real world clinical experience. A major reason for the high morbidity and mortality is that the heart has an inadequate regenerative response to the myocardial necrosis sustained following AMI; cell death from the ischemic damage can lead to progressive ventricular dilation and dysfunction through the processes of adverse left ventricular remodelling. However, the discovery of tissue resident cardiac stem cells in the mammalian heart [5] has challenged the long held belief that the heart is a terminally-differentiated organ and opens up the possibility of using bone marrow derived stem cells to repair the heart. Indeed, recent experimental studies documented that bone marrow-derived cell (BMC) injection into the infarcted heart stimulates the formation of newly formed cardiac myocytes, although the origin of these myocytes is still a matter of debate[6]. Numerous pre-clinical studies provided high degree of evidence that bone marrow derived cells do contribute to cardiac repair after acute myocardial injury, limit infarct expansion and improve cardiac function most likely via a paracrine mechanism of action. Pre-clinical evidence is corroborated by several small to intermediate size clinical trials demonstrating beneficial effects of bone marrow derived cells on top of the state-of-the-art reperfusion treatment [7]. For this reason, European Community has recently funded within FP-7 "The effect of intracoronary reinfusion of bone marrow derived mononuclear cells (BM-MNC) on all cause-mortality in acute myocardial infarction (BAMI)" project aimed to definitively demonstrate the efficacy of BM-MNC in patients with myocardial infarction.

   Considering that recovery of post-infarction LV function is favourably correlated to bone marrow derived stem cell mobilization induced by endogenous Granulocyte-Colony Stimulating Factor (G-CSF) [8-9], therapeutic stem cell mobilization was proposed as an alternative method to ameliorate post-infarction LV function. Several basic studies have supported this notion suggesting that stem cell mobilization might improve LV function by increasing stem cell homing in the damaged myocardium in addition to a favourable direct effect of G-CSF on LV myocardium [10-12].

   On these bases several studies have evaluated the effect of G-CSF on LV function in patients with myocardial result with mixed results [13]. In general, G-CSF was proven safe but the effect appeared modest. However, in patients with large myocardial infarction the effect was significant and clinically relevant approaching a 5% increase in LVEF. In particular in the Rigenera Trial conducted at the Catholic University of the Sacred Heart of Rome 41 patients with large anterior wall AMI at high risk of unfavorable remodeling were randomized 1:2 to Lenograstim (rhu G-CSF, Myelostim 34, Italfarmaco) (10 μg/kg/day for 5 days) or to conventional therapy. After a median follow-up of 5 months patients treated with Lenograstim exhibited improvement of 5% in LVEF, in the absence of LV dilation. In contrast, patients treated conventionally exhibited significant LV dilation in the absence of an improvement in LVEF [14]. In the present study, a subgroup of 8 patients randomized to Lenograstim received also the administration of a second-generation ultrasound contrast agent containing sulphur hexafluoride (SonoVue®, Bracco, Milan, Italy) administered intravenously (5 ml at 1 ml/min) for myocardial opacification to collect diagnostic images by Myocardial Contrast Echocardiography. Interestingly, a post hoc analysis, revealed that only patients receiving Sonovue® showed a significant benefit on LV function [unpublished data]. This could be due to an increased homing effect of mobilized bone marrow derived stem cells due to the myocardial destruction of contrast medium-microbubbles by 3.5 MHz ultrasounds produced by the Echo machine. As this regard, two basic studies demonstrated that the highly focused ultrasound-mediated stimulation of microbubbles increased the migration of stem cells across the myocardial endothelium into the post-ischemic myocardium in vivo [15-16]. Moreover, long term (10 years) follow up data of the RIGENERA trial have been recently collected, confirming the safety of the procedure and a significant improvement of the quality of life assessed by NYHA functional class, Seattle Heart Failure Model, Minnesota Living with Heart Failure Questionnaire (p<0.005) when compairing patients treated with G-CSF versus standard therapy. Data regarding efficacy, in terms of LVEF, end-diastolic volume and end-systolic volume are currently under analysis.

   On the basis of the previous results, The Recupero dall'Infarto miocardico con G-CSF E Nuovi Esempi di Rigenerazione Avanzata (RIGENERA 2.0) trial will specifically test the efficacy of the combined effect of subcutaneous Granulocyte - Colony Stimulating Factor and sulphur hexafluoride on post-infarction left ventricular function.

   1.2 BENEFIT-RISK ASSESSMENT In every clinical trial, anticipated benefits need to be weighed against the study associated risks. In previous investigations where G-CSF has been used, no G-CSF associated adverse reactions were reported. Only the MAGIC trial was prematurely stopped due to possible safety concerns in treated patients in terms of an unexpectedly high restenosis rate in stented vessels [17]. However, only three patients in the G-CSF group received angiographic follow-up, thus no clear conclusion about the incidence of restenosis should have reasonably be drawn from this study. In all other studies using G-CSF adverse events were comparable between patients and controls [13]. Nevertheless G-CSF is largely used in oncology for treatment of febrile neutropenia and in hematology for this indication and for mobilization of stem cells for transplantation. As this regard G-CSF is considered reasonably safe without any association with a documented increase in malignancies [18].

   SonoVue has been shown to be safe and well tolerated with minimal risk to patients. In clinical trials, the overall incidence of adverse events was relatively low (10.7% overall, 5.2% investigational product-related) in subjects receiving SonoVue. The most frequently reported adverse events were headache (2.1%), nausea (0.9%), chest pain (0.8%), and chest discomfort (0.5%). All other adverse events occurred at a frequency of <0.5%. Most adverse events were mild and resolved spontaneously within a short time without sequelae. Serious adverse events occurred in 0.43% of patients and only 0.08% of events were considered to be of some relationship to the administration of SonoVue (probable, possible, or unlikely). No product- related deaths were reported within MAH-sponsored trials.

   The anticipated benefits of RIGENERA 2.0 trial for study participants are expected better LV function, a parameter that is well-known to influence long-term outcome. Nevertheless, chiefs of the different Units involved in the present study will form a Data Monitoring Committee that will stop the study in case of an observed increase in the rate of adverse events.
2. STUDY OBJECTIVES 2.1. PRIMARY OBJECTIVE Primary efficacy endpoint

   • Left ventricular ejection fraction (LVEF) at 6 months assessed by Cardiac Magnetic Resonance and centrally reviewed

   Secondary efficacy endpoints:
   * Left ventricular end-diastolic volume (LVEDV) assessed by Cardiac Magnetic Resonance at 6 months at 6 months and centrally reviewed
   * Left ventricular end-systolic volume (LVEDV) assessed by Cardiac Magnetic Resonance at 6 months and centrally reviewed
   * Left ventricular ejection fraction (LVEF) assessed by 2D Echocardiography at 6 months and centrally reviewed
   * Left ventricular end-diastolic volume (LVEDV) assessed by 2D Echocardiography at 6 months and centrally reviewed
   * Left ventricular end-systolic volume (LVEDV) assessed by 2D Echocardiography at 6 months and centrally reviewed
   * Incidence of clinical major adverse events (death, myocardial infarction, sustained cardiac arrhythmias, cardiogenic shock, stroke and rehospitalization due to heart failure at 1 year).

   Safety endpoints:

   • Incidence of new neoplastic and hematological diseases
3. OVERALL DESIGN AND PLAN OF THE STUDY 3.1. OVERVIEW OF STUDY FLOW The RIGENERA 2.0 trial is a phase II placebo-controlled, randomized, open label, with Blinded Evaluation of end-points. One hundred and twenty STEMI patients are planned to be enrolled in 4 Italian centers (Rome - Catholic University of the Sacred Heart, Ferrara, Pisa and Padua). Patients with an acute ST-elevation myocardial infarction as defined by the universal definition of AMI undergoing acute revascularization (i.e. either acute PCI within 24 hours of symptom onset or thrombolysis within 12 hours followed by acute PCI within 24 hours of symptom onset) will be screened at investigational sites. Patients who had acute PCI at institutions different from the investigational sites (recruiting centers) can also be included: interested patients may be referred for screening to any of the participating study sites within 3 to 4 days. Informed consent and assessment of eligibility of patients with respect to in- and exclusion criteria will be done at the recruiting centers. If all other eligibility criteria are met, echocardiography will be performed 3 to 6 days after the acute PCI and ejection fraction will be quantified. In case of LVEF≤45% the patient will be 1:1 electronically randomized to G-CSF and MCE or placebo and MCE according to site. Patients will be randomized to receive either subcutaneous Granulocyte - Colony Stimulating Factor (group 1) or Placebo (group 2) both added on top of optimal standard of care and Myocardial Contrast Echocardiography with intravenous infusion of sulphur hexafluoride.

Lenograstim (rhu G-CSF, Myelostim 34, Italfarmaco) (5 µg/kg twice daily for 5 days, subcutaneously) or placebo (saline solution twice daily for 5 days, subcutaneously) will be administered at least 5 days after admission.

Both in patients treated with Lenograstim (rhu G-CSF, Myelostim 34, Italfarmaco) and in patients treated with placebo, immediately before the first dose of Lenograstim (rhu G-CSF, Myelostim 34, Italfarmaco) or placebo and in the morning of the last day of treatment in which the peak of BMSC mobilization is expected, an echocardiogram using an echocardiographic contrast agent (Sonovue, Bracco) will be performed. In the days of administration of the drug or placebo, ECG, blood pressure, blood count and coagulation analyses will be monitored.

In the case of muscle and bone pain or severe headache patients will be treated with paracetamol.

In the case of leukocytosis (> 40000/mcl) dose of G-CSF in 24 hours will be halved and in the case of leukocytosis (> 70000/mcl) completely stopped.

After hospital discharge, all study patients will return to the clinical centre for a follow up visit after 30 days. Six months after randomization all the patients will undergo outpatient Cardiac Magnetic Resonance and Conventional Echocardiography. At the same time, all patients will undergo Myocardial Contrast Echocardiography. At 1 year all patients will attend a final site visit at the clinical centers collecting any clinical event. However, all clinical endpoints will be reported as occurring throughout the follow up. Clinical Major adverse cardio-cerebrovascular events (death, myocardial infarction, stroke and re-hospitalization due to heart failure) at 1 year will be adjudicated by a clinical event committee blinded to the patient treatment allocation. This will ensure a consistent and unbiased adjudication of events across all investigational sites.

3.2. STUDY POPULATION 3.2.1. Number of patients A total of approximately 120 male and female patients are planned to be enrolled in the RIGENERA 2.0 trial. Enrolment will involve 4 Italian centres (Roma, Pisa, Ferrara, Padua). Recruiting centres will keep a log of all patients proposed to be included.

3.2.2. Inclusion criteria

1. Signed and dated informed consent
2. Men and women of any ethnic origin aged ≥ 18 years
3. Patients with acute ST-elevation myocardial infarction as defined by the universal definition of AMI.
4. Successful acute reperfusion therapy (residual stenosis visually <50% and TIMI flow ≥2) within 24 hours of symptom onset or thrombolysis within 12 hours of symptom onset followed by successful percutaneous coronary intervention (PCI) within 24 hours after thrombolysis
5. Left ventricular ejection fraction ≤ 45% with significant regional wall motion abnormality assessed by quantitative echocardiography 3 to 6 days after reperfusion therapy

3.3.3. Exclusion criteria

1. Participation in another clinical trial within 30 days prior to randomization
2. Pregnant or nursing women or women in childbearing age not able to esclude the possibility of a pregnancy
3. Mental condition rendering the patient unable to understand the nature, scope and possible consequences of the study or to follow the protocol
4. Necessity to revascularize additional vessels, outside the target coronary artery after investigational therapy/placebo administration (additional revascularizations after primary PCI and before investigational therapy/placebo administration are allowed)
5. Persistent cardiogenic shock
6. Known hematologic and neoplastic diseases
7. Severe impaired renal function, i.e. eGFR<30 ml/min
8. Persistent fever or diarrhoea not responsive to treatment within 4 weeks prior screening or severe infection
9. Uncontrolled hypertension (systolic >180 mmHg and diastolic >120 mmHg)
10. Life expectancy of less than 2 years from any non-cardiac cause or neoplastic disease

4. STUDY CONDUCT 4.1. SCHEDULE OF PROCEDURES The schedule of study assessment is listed in Table 1. Screening Days -6 to - 3 Randomization Treatment Day 0 to 5 Recovery Day 5 to 10 1 month 4-6 Months Informed Consent X Demographics X Medical History X Killip Class X X X NYHA Class X X X Physical Examination X X X Vital Signs (BP and HR) X X X ECG X X X Safety Laboratory X X (daily) X X X Concomitant Medications X X X Adverse Event / Endpoint Collection X X X X Echocardiography+ X X Magnetic Resonance X X Recommended but optional Bloods (see below) X X X Urine Pregnancy test(where applicable) X X X Investigational therapy X X

♦Recommended but optional Bloods Screening:

Hematology: Red blood count, white blood count Biochemistry and enzymes: serum urea, serum uric acid, glutamic-oxaloacetic transaminase (GOT), glutamic-pyruvate transaminase (GPT), lactate dehydrogenase (LDH), total cholesterol, low density lipoprotein cholesterol (LDL), high density lipoprotein cholesterol (HDL), triglycerides, glycosylated hemoglobin (HbA1c) Electrolytes: sodium, potassium Cardiac marker: Creatine kinase (CK), Creatine kinase muscle-brain (CK-MB), (high sensitive) troponin T or I Coagulation: International Normalised Ratio (INR) Hematology: hemoglobin, hematocrit, red blood count, white blood count, platelets Biochemistry and enzymes: serum urea, serum uric acid, GOT, GPT, LDH, total cholesterol, LDL-cholesterol., HDL-cholesterol, triglycerides, HbA1C Electrolytes: sodium, potassium Cardiac marker: CK, CK-MB, (high sensitive) troponin T or I Coagulation: INR

4.2. PATIENT SCREENING AND RANDOMISATION Patients will be recruited based on the existing medical information from the pool of AMI patients at the clinical centres. Patients who had the primary PCI performed at clinical centres that are different from the recruiting centre can also be included: interested patients may be referred for screening to any of the participating study sites within 3 to 4 days. Informed consent and assessment of eligibility of patients with respect to inclusion and exclusion criteria will be done at the recruiting centre. Written informed consent must be obtained from patients prior to any study specific procedures. After consenting, patients undergo the procedures listed for the screening visit. After ensuring that a patient meets all other eligibility criteria, the investigator will perform the echocardiography and an electronic record of the echocardiography will be kept and transferred to the central Echocardiography Core Laboratory for following analyses. After local quantification of left ventricular ejection fraction, randomisation will be allowed for all patients with LVEF ≤ 45%. At randomization a patient number that will be used as the key identifier for the entire study period, will be supplied. Patients will be randomised to investigational therapy or placebo in a 1:1 ratio. Patients with a LVEF > 45% will not be randomised, but will be classified as screening failures. Patients randomised but not treated will be replaced. Patients who discontinue the study after treatment, will not be replaced.

4.3. DESCRIPTION OF STUDY ASSESSMENTS 4.3.1. Medical history / demographics A complete medical history will be obtained from each patient at the screening visit. Demographics, including gender, age and ethnic origin, and the smoking status will be recorded.

4.3.2. Killip Class

Patients will be ranked according to the Killip Class status. Definitions of the grading system are as follows:

Class I: Absence of rales over the lung fields and absence of S3. No heart failure. No clinical signs of decompensation.

Class II: Rales over 50% or less of the lung fields or the presence of an S3. Heart failure. Diagnostic criteria include rales, S3 gallop and venous hypertension.

Class III: Rales over more than 50% of the lung fields. Severe heart failure. Frank pulmonary edema.

Class IV: Cardiogenic shock. Hypotension (a systolic blood pressure of less than 90 mmHg for at least 30 minutes or the need for supportive measures to maintain a systolic blood pressure of greater than or equal to 90 mmHg), end-organ hypoperfusion (cool extremities or a urine output of less than 30 ml/h, and a heart rate of greater than or equal to 60 beats per minute). The hemodynamic criteria are a cardiac index of no more than 2.2 l/min per square meter of body-surface area and a pulmonary capillary wedge pressure of at least 15 mmHg. Signs include hypotension (systolic pressure < 90 mm Hg) and evidence of peripheral vasoconstriction such as oliguria, cyanosis and diaphoresis. Heart failure, often with pulmonary oedema, has also been present in the majority of these patients.

4.3.3. Physical examination All patients will undergo standard or abbreviated physical examinations. The standard examination is based on the following body systems: body temperature, HEENT (head, eyes, ears, nose, throat), respiratory system, cardiovascular system, abdomen, extremities, neurological system. The abbreviated physical examination consists of body temperature, respiratory system, cardiovascular system, and lymph nodes. The body weight will be determined at each physical examination. The body height will be obtained at screening only.

4.3.4. Vital signs Blood pressure and heart rate at rest will be determined using a standard method.

4.3.5. Electrocardiography A 12 lead electrocardiogram (ECG) will be recorded. ECGs will be recorded while the patient is resting in supine position. Abnormal findings in ECG recordings will be documented and the clinical relevance will be judged. A de-identified copy of the baseline ECG will be digitally stored.

4.3.6. Clinical laboratory Blood sampling and sample analysis will be performed at the clinical centre. The local investigator is responsible for proper judgment of abnormal blood test results, and is responsible for appropriate patient care following clinically significant pathological results. Please refer to section 6.4.5 to determine whether an abnormal laboratory value may constitute an adverse event.

The following analysis will be obtained at screening, daily during the five days of treatment (from day 0 to day 5) and at 5, 30 and 180 days:

Screening:

Hematology: Hemoglobin, hematocrit, Red blood count, white blood count, platelets Biochemistry: Serum creatinine, serum urea, serum uric acid, glutamic-oxaloacetic transaminase (GOT), glutamic-pyruvate transaminase (GPT), lactate dehydrogenase (LDH), total cholesterol, low density lipoprotein cholesterol (LDL), high density lipoprotein cholesterol (HDL), triglycerides, glycosylated hemoglobin(HbA1c), Creatine kinase (CK), Creatine kinase muscle-brain(CK-MB), high sensitive troponin T hs-TnT, Vascular Endothelial Growth Factor (VEGF), Insulin Growth Factor 1 (IGF-1), hepatocyte Growth Factor (HGF), Stromal Derived Factor 1 alpha (SDF-1 alpha) Urine: Pregnancy test for woman of childbearing potential Coagulation: Prothrombin Time (PT), International Normalised Ratio (INR), activated partial thromboplastin time (aPTT) 4.3.7. Concomitant medications All patients participating in the trial should receive treatment according to evidence based guidelines. Concomitant medications will be recorded throughout the study.

4.3.8. Standard Echocardiography A resting echocardiogram at enrollment and at 4-6 months will be recorded and digitally stored. See details in 5.3.1 Only if the patient qualifies with LVEF ≤ 45% in the local reading, the patients will be randomised

4.3.9. Investigational therapy/placebo Lenograstim (rhu G-CSF, Myelostim 34, Italfarmaco) (5 µg/kg twice daily for 5 days, subcutaneously) or placebo (saline solution twice daily for 5 days, subcutaneously) will be administered at least 5 days after admission.

Both in patients treated with Lenograstim (rhu G-CSF, Myelostim 34, Italfarmaco) and in patients treated with placebo, immediately before the first dose of Lenograstim (rhu G-CSF, Myelostim 34, Italfarmaco) or placebo and in the morning of the last day of treatment in which the peak of BMSC mobilization is expected, an echocardiogram using an echocardiographic contrast agent (Sonovue, Bracco) will be performed in the days of administration of the drug or placebo, ECG, blood pressure, blood count and coagulation analyses will be monitored.

In the case of muscle and bone pain or severe headache patients will be treated with paracetamol.

In the case of leukocytosis (> 40000/mcl) dose of G-CSF in 24 hours will be halved and in the case of leukocytosis (> 70000/mcl) completely stopped.

Patients will be safely discharged on the basis of laboratory data.

4.4. DURATION OF THE STUDY 4.4.1. Study duration for study patients Each enrolled patient will remain in the study throughout the entire study duration, with a minimum follow-up of 1 year for each patient. A study patient's participation may be terminated early for reasonable cause, such as the investigator's medical decision. At any time, the patient has the right to withdraw consent without a negative impact on her/his medical treatment. However, the investigators are encouraged to ask for the patient's permission for further follow-up telephone contacts from those whose decision for discontinuation was based on the need for further outpatient visits.

4.4.2. Duration of the whole study Patients will be enrolled during a recruitment phase of approximately 2 years. Since minimum study duration for one patient is one year, the overall study duration is approximately 3 years. The Data Monitoring Committee may terminate the study earlier based on safety concerns at any time, or based on the interim efficacy analysis. Competent authorities/ethics committees retain the right for premature termination of the study according to applicable regulations. At an individual study centre, the study may be terminated early if the work performed is not compliant with Good Clinical Practice (GCP).

ELIGIBILITY:
Population Adult male or female patients aged < 80 years with acute myocardial infarction undergoing successful primary or rescue percutaneous recanalization of the infarct-related coronary artery, defined as TIMI 3 flow and residual stenosis <20%) within 24 hours of symptom onset and Left Ventricular Ejection Fraction (LVEF) ≤ 45% at 3-6 after revascularization, as documented by a two-dimensional echocardiogram.

Inclusion Criteria:

1. Signed and dated informed consent
2. Men and women of any ethnic origin aged ≥ 18 years
3. Patients with acute ST-elevation myocardial infarction as defined by the universal definition of AMI.
4. Successful acute reperfusion therapy (residual stenosis visually <50% and TIMI flow ≥2) within 24 hours of symptom onset by successful percutaneous coronary intervention (PCI) or thrombolysis within 12 hours of symptom onset followed by successful PCI within 24 hours after thrombolysis
5. Left ventricular ejection fraction ≤ 45% at 24 hours after revascularization, as documented by a two-dimensional echocardiogram.

Exclusion Criteria:

1. Participation in another clinical trial within 30 days prior to randomisation
2. Pregnant or nursing women or women in childbearing age not able to esclude the possibility of a pregnancy
3. Mental condition rendering the patient unable to understand the nature, scope and possible consequences of the study or to follow the protocol
4. Necessity to revascularise additional vessels, outside the target coronary artery after investigational therapy/placebo administration (additional revascularisations after primary PCI and before investigational therapy/placebo administration are allowed)
5. Persistent cardiogenic shock
6. Known hematologic and neoplastic diseases
7. Severe impaired renal function, i.e. GFR<30 ml/min
8. Persistent fever or diarrhoea not responsive to treatment within 4 weeks prior screening or severe infection
9. Uncontrolled hypertension (systolic >180 mmHg and diastolic >120 mmHg)
10. Life expectancy of less than 2 years from any non-cardiac cause or neoplastic disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-01 (Estimated); Primary Completion 2021-10 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Left ventricular ejection Fraction | 6 months
  Left ventricular ejection fraction (LVEF) at 6 months assessed by Cardiac Magnetic Resonance and centrally reviewed

SECONDARY OUTCOMES:
Left ventricular end-diastolic volume (LVEDV) | 6 months
  Left ventricular end-diastolic volume (LVEDV) assessed by Cardiac Magnetic Resonance at 6 months and centrally reviewed
Left ventricular end-systolic volume (LVEDV) | 6 months
  Left ventricular end-systolic volume (LVEDV) assessed by Cardiac Magnetic Resonance at 6 months and centrally reviewed
Left ventricular ejection fraction (LVEF) | 6 months
  Left ventricular ejection fraction (LVEF) assessed by 2D Echocardiography at 6 months and centrally reviewed
Left ventricular end-diastolic volume (LVEDV) | 6 months
  Left ventricular end-diastolic volume (LVEDV) assessed by 2D Echocardiography at 6 months and centrally reviewed
Left ventricular end-systolic volume (LVESV) | 6 months
  Left ventricular end-systolic volume (LVEDV) assessed by 2D Echocardiography at 6 months and centrally reviewed
MACCE | 1 year
  Clinical Major adverse cardio-cerebrovascular events (death, myocardial infarction, stroke and rehospitalization due to heart failure) at 1 year

OTHER OUTCOMES:
Incidence of adverse events | 1 years
  adverse events
Incidence of new neoplastic and hematological diseases | 5 years
  neoplastic and hematological diseases

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Maria Leone, MD, PhD, Principal Investigator — Universita' Cattolica del Sacro Cuore; Filippo Crea, MD, Study Chair — Universita' Cattolica del Sacro Cuore
Locations (1):
- Fondazione Policlinico Universitario Agostino Gemelli, Rome, RM, Italy

REFERENCES:
- [Derived] Leone AM, D'Amario D, Teofili L, Basile E, Cannata F, Graziani F, Marzilli M, Russo AM, Tarantini G, Ceconi C, Leone G, Trani C, Rebuzzi AG, Crea F. The combined effect of subcutaneous granulocyte- colony stimulating factor and myocardial contrast echocardiography with intravenous infusion of sulfur hexafluoride on post-infarction left ventricular function, the RIGENERA 2.0 trial: study protocol for a randomized controlled trial. Trials. 2016 Feb 19;17:97. doi: 10.1186/s13063-016-1172-0. PMID 26891753